CLINICAL TRIAL: NCT04499352
Title: An Open Label, Randomized Phase II Study of BI 754091 Alone or in Combination With BI 836880 in Patients With Chemotherapy Resistant, Unresectable, Metastatic Squamous Cell Carcinoma of the Anal Canal
Brief Title: A Study to Test BI 754091 Alone or in Combination With BI 836880 in People Who Have Advanced Anal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Not due to safety reasons (sponsor decision).
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1381-0011; 2019-004749-33 (EudraCT Number)
Record Dates: First submitted 2020-08-03; First posted 2020-08-05 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Anal Canal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- treatment arm A (Experimental)
  Interventions: Drug: BI 754091
- treatment arm B (Experimental)
  Interventions: Drug: BI 754091; Drug: BI 836880

INTERVENTIONS:
Drug: BI 754091 — BI 754091
Drug: BI 836880 — BI 836880
  Arms: treatment arm B

SUMMARY:
The objective of this trial is to assess anti-tumour activity of BI 754091 as monotherapy and of BI 754091 in combination with BI 836880 in patients with unresectable or metastatic squamous cell carcinoma of the anal canal who progressed on or after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written Informed Consent Form (ICF) in accordance with ICH-GCP and local legislation prior to admission to the trial.
2. Patients ≥18 years of age or over the legal age of consent in countries where that is greater than 18 years at the time of signature of the ICF.
3. Patients must have histologically or cytologically documented surgically unresectable locally-advanced or metastatic Squamous cell carcinoma of the anal canal (SCCA).
4. Patients with loco-regional anal cancer as initial diagnosis must have unresectable progressive locally advanced or metastatic SCCA after failure of at least one line (but not more than two lines) of previous systemic treatment unless ineligible for or intolerant to this systemic therapy.

   Patients with metastatic anal cancer as initial diagnosis (no prior treatment for loco-regional cancer) must have failed one line of previous systemic treatment (chemotherapy ± radiotherapy) for the metastatic anal cancer unless ineligible for or intolerant to this systemic treatment. (Patients with metastatic anal cancer as initial diagnosis who have received two or more lines of systemic treatment for the metastatic anal cancer are not eligible for the study.)
5. All patients must have at least one measurable lesion according to RECIST v1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status score 0 to 1
7. All patients must be willing to undergo blood testing for human immunodeficiency virus (HIV) presence in the blood if not tested within the past 6 months prior to signature of ICF for this trial.

   For patients confirmed as HIV positive, all of the following (a-d) applies:
   1. CD4+ count ≥ 250 cells/μL
   2. Undetectable viral load (local lab assessment)
   3. Must be currently receiving Highly Active Antiretroviral Therapy
   4. A HIV/Infectious Diseases specialist must be consulted or patient must be under the care of the HIV/Infectious Diseases specialist
8. Patients must be willing to allow programmed cell death ligand 1 (PD-L1) status assessment by one of following options.

   Preference is given to fresh tumour biopsy sample collection at baseline before receiving first trial medication. In case a fresh tumour biopsy cannot be obtained (e.g. inaccessible lesions or patient safety concern), archival tissue will be requested. If neither is available any previous historical information regarding PD-L1 status should be collected via eCRF. Exceptions may be considered after consultation with and approval by the Sponsor.
9. Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, for the entire duration of the trial treatment intake and for 6 months after the end of the trial treatment. A list of contraception methods meeting these criteria is provided in the patient information.

Exclusion Criteria:

1. Current or prior treatment with any systemic anti-cancer therapy or any investigational product (or device) either within 28 days or less than 5 half-lives (whichever is shorter) before start of trial treatment.
2. Major injuries and/or surgery or bone fracture within 4 weeks of start of treatment, or planned surgical procedures during the trial period.
3. Significant cardiovascular/cerebrovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 6 months, congestive heart failure > New York Heart Association (NYHA) II).

   Uncontrolled hypertension is defined as: blood pressure in rested and relaxed condition ≥ 140 mmHg, systolic or ≥ 90 mmHg diastolic (with or without medication)
4. Known inherited predisposition to bleeding or to thrombosis in the opinion of the investigator.
5. History of severe hemorrhagic or thromboembolic event in the past 12 months (excluding central venous catheter thrombosis and peripheral deep vein thrombosis).
6. Patients who require full-dose anticoagulation (according to local guidelines). No Vitamin K antagonist and other anticoagulation allowed; Low-Molecular-Weight-Heparin (LMWH) and acetylsalicylic acid (ASA) allowed only for prevention not for curative treatment.
7. Prior treatment with anti-PD-1, anti-PD-L1, or anti CTLA-4 treatment
8. Prior treatment with any antiangiogenic agent (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL-184, sunitinib, etc.) Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Objective response (OR) | up to 3 years

SECONDARY OUTCOMES:
Duration of objective response (DoR) | up to 3 years
Progression-free survival (PFS) | up to 3 years
Overall survival (OS) | up to 3 years
Disease control (DC) | up to 3 years
Adverse events (AEs) | up to 3 years
Drug related AEs from the time of treatment initiation until the end of the Residual Effect Period (REP) | up to 3 years
Drug related AEs leading to dose reduction of BI 836880 and/or discontinuation of study treatment (i.e. both trial drugs) | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com